CLINICAL TRIAL: NCT02854163
Title: An Exploration of the Dynamic Interaction Between IL-17, IL-17 Inhibition With (Secukinumab) and Neutrophils in Psoriatic Arthritis in Vitro and ex Vivo With Exploratory Study on the Potential Role of Vitamin D
Brief Title: Effect of Secukinumab in the Treatment of Psoriatic Arthritis
Acronym: SATURN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Robert J Moots, Professor of Rheumatology, University of Liverpool
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UoL001145; 2015-004502-42 (EudraCT Number); LCTU134 (Other: Cancer Research UK LCTU, Liverpool); CAIN457F2208T (Other Grant/Funding Number: NOVARTIS)
Record Dates: First submitted 2016-07-20; First posted 2016-08-03 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Psoriatic Arthritis
Keywords: Secukinumab; Neutrophils; Vitamin D
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Secukinumab (Experimental): Secukinumab will be given to all 20 patients registered (Secukinumab group). All doses will be given subcutaneously using the following schedule: 4 weekly injections of 150 or 300 mg subcutaneous injections depending the severity of skin involvement, followed by 11 monthly subcutaneous injections of 150mg.
  Patients will continue to use their normal DMARDs treatment.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — All eligible patients registered into the study will receive four 150 - 300 mg subcutaneous injections at weekly intervals, followed by regular injections 150mg once a month thereafter for a total of 12 months
  Other Names: Cosentyx

SUMMARY:
The investigators propose an open label pragmatic clinical and laboratory study designed to investigate, in detail, the clinical and molecular effects of Interleukin 17 (IL-17) and inhibition of IL-17 with secukinumab, on neutrophil function in vitro and ex vivo.

As secondary, exploratory objectives, the investigators will utilise the fact that secukinumab is to be administering to 20 patients with Psoriatic Arthritis (PsA) and investigate whether there is any relationship between vitamin D status and response to secukinumab, with respect to efficacy and adverse events. The results of this secondary exploratory analysis will inform the design of a larger, definitive study.

DETAILED DESCRIPTION:
Phase: Phase 2 Clinical Trial of an Investigational Medicinal Product (CTIMP)

Sample Size: 20 patients plus 10 healthy controls are to be enrolled in total.

Study Population:

Patient treatment group: 20 patients with active psoriatic arthritis (fulfilling Classification Criteria for Psoriatic Arthritis [CASPAR] criteria) affecting ≥2 peripheral joints (swollen and tender) that have not responded to at least one standard Disease-modifying antirheumatic drugs (DMARDs).

Healthy control group: 10 healthy control blood samples (matched for gender to the patients and within 5 years of mean age within each gender subgroup).

Number of Sites: 1 - Rheumatology clinic at Aintree University Hospital, Liverpool

Study Duration: 24 months in total with 12 months of therapy, and 12 months for staggered enrolment and laboratory investigations

Description of Agent/Intervention

Secukinumab 150mg/300mg subcutaneous injection once weekly for the first 4 weeks then 150mg subcutaneous injection 4 weekly for up to 11 months.

Primary Aim:

The primary aim is to determine the molecular effects of IL-17 and inhibition of IL-17 with secukinumab on neutrophil phenotype, lifespan, function and production of IL-17.

Secondary Aims:

1. To determine if neutrophil life span and function is associated with vitamin D concentration and VDR receptor expression in PsA patients, and
2. To explore whether vitamin D concentrations and VDR expression influence neutrophil lifespan and function in PsA patients before and after treatment with secukinumab.

Exploratory Aims:

1. To evaluate the clinical response of patients with psoriatic arthritis, treated with secukinumab using Psoriasis Area and Severity Index (PASI 75) and American College of Rheumatology response criteria (ACR20),
2. To identify whether vitamin D status according to winter or summer seasons and levels of VDR expression are associated with skin and joint responses or infection in patients treated with secukinumab in PsA, assessed using PASI 75 and 90, ACR20 response and reporting of infection adverse events.
3. To evaluate the safety of patients treated with secukinumab in terms of adverse events (AE), serious adverse events (SAE), infections and serious infections, malignancies, acute injection site reactions and potential immunogenicity over 12 months.

Study Design:

Screening for eligibility

Patient group: Patients attending routine rheumatology assessments will be screened for suitability for the study. Eligible patients, based on diagnosis of PsA (meeting CASPAR criteria and with peripheral joint involvement), will be approached to determine if they are willing to participate.

Eligible patients will be registered into the study and will receive secukinumab treatment in addition to their standard DMARD treatment.

Healthy Control Group: Healthy controls matched by gender and within 5 years of mean patient age (assessed in patient group) will be recruited from National health Service (NHS) and university staff.

Baseline assessment:

Baseline assessment of Vitamin D, VDR, Neutrophil function ACR20, Body Surface Area (BSA), PASI 75 and 90, Nail Psoriasis Severity Index (NAPSI), Psoriatic Arthritis Response Criteria (PSARC), EuroQol five dimensions questionnaire (EQ5D) & Health Assessment Questionnaire (HAQ).

1. Secukinumab group

   3 months - assessment of Vitamin D, VDR, Neutrophil function, ACR20, PASI 75 AND 90, NAPSI, PSARC, EQ5D, HAQ

   6 months - assessment of Vitamin D, VDR, Neutrophil function, ACR20, PASI 75 AND 90, NAPSI, PSARC, EQ5D, HAQ

   9 months - assessment of Vitamin D, VDR , ACR20, PASI 75 AND 90, NAPSI, PSARC, EQ5D HAQ

   12 months - assessment of Vitamin D, VDR, Neutrophil function, ACR20, PASI 75 AND 90, NAPSI, PSARC, EQ5D, HAQ

   13 months (final follow up visit) - pregnancy test, Full Blood Count (FBC), LFTs, serum creatinine and body temperature measurement.

   Then exit study
2. Healthy Control Group: Blood sample obtained at baseline for assessment of Vitamin D, VDR and neutrophil function.

Analysis Plan:

Phase 1:

* Measure change at 3 month, 6 and 12 months assessments (from baseline) in neutrophil function, in the secukinumab group.

Phase 2:

* Measure vitamin D concentration, VDR at 3 months, 6 months, 9 months and 12 months.
* Model fluctuation in vitamin D, which is season dependant and estimate when it is maximal.
* Compare treatment response at time point treatment with lowest vitamin D concentration (winter time) with that with highest vitamin D concentration (summer time).
* Assess whether difference in neutrophil function, ACR20, PASI 75 and 90 response and NAPSI correlate with change in vitamin D, using longitudinal models

ELIGIBILITY:
Patients Inclusion Criteria:

* Patients with active psoriatic arthritis (fulfilling CASPAR criteria) affecting ≥2 peripheral joints (swollen and tender) that have not responded to at least one standard DMARDs
* All meet CASPAR criteria for diagnosis of PsA,
* Be rheumatoid factor and anti-cyclic citrullinated peptide (anti-CCP) negative at screening,
* Have had no prior exposure to biologic therapy,
* Not have received parenteral glucocorticosteroids in the 6 weeks prior to the baseline assessment,
* If taking oral glucocorticoids remain on a stable dose of <10mg throughout the study with no change in dose in the 6 weeks prior to baseline assessment,
* If taking methotrexate or other DMARDs remain on a stable dose throughout the study and not have changed dose or therapy for 6 weeks prior to the baseline assessment

Patients Exclusion Criteria:

* Active or chronic infection including mycobacterium tuberculosis, HIV, hepatitis B or C
* Absence of active psoriatic arthritis
* Patients who are starting anti-TNF therapy for treating PsA
* Pregnancy and planning pregnancy

  1. WOCBP who are unwilling or unable ot use acceptable method to avoid pregnancy for study duration plus timeframe as specified in section 5.2.5.
  2. Women who are pregnant or breastfeeding
  3. Sexually active fertile men not using effective birth control if their partners are WOCBP.
* Malignancy
* Chest X-ray or chest MRI with evidence of ongoing infectious or malignant process obtained within 3 months prior to Screening and evaluated by a qualified physician.
* Patients with hyponatraemia and nephrotic syndrome
* Previous exposure to secukinumab or other biologic drug directly targeting IL-17 or IL-17 receptor.
* Use of any investigational drug and/or devices within 4 weeks before registration or a period of 5 half-lives of the investigational drug, whichever is longer.
* Significant comorbidity that, in the opinion of the investigator, would impact on ability to participate
* Any change in the dose of oral glucocorticosteroids or DMARDS in the prior 6 weeks prior to the Baseline visit or use of i.v. intramuscular or intra-articular glucocorticosteroid during the last 6 weeks prior to the enrolment visit.
* Patients who have previously been treated with TNFα inhibitors (investigational or approved).
* History of hypersensitivity to the study drug or its excipients or to drugs of similar classes.
* Previous treatment with any cell-depleting therapies including but not limited to anti-CD20 investigational agents (e.g. CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19).
* Active ongoing inflammatory diseases other than PsA that might confound the evaluation of the benefit of secukinumab therapy.
* Underlying metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine,cardiac, infectious or gastrointestinal conditions which in the opinion of the Investigator immunocompromise the patient and/or place the patient at unacceptable risk for participation in an immunomodulatory therapy.
* Significant medical problems or diseases, including but not limited to the following: uncontrolled hypertension (≥ 160/95 mmHg), congestive heart failure (New York Heart Association status of class III or IV), uncontrolled diabetes.
* History of clinically significant liver disease or liver injury as indicated by abnormal liver function tests (LFT) such as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, or serum bilirubin. The Investigator should be guided by the following criteria:

  1. Any single parameter may not exceed 2 x upper limit of normal (ULN). A single parameter elevated up to and including 2 x ULN should be re-checked once more as soon as possible, and in all cases, at least prior to enrollment/registration, to rule out laboratory error.
  2. If the total bilirubin concentration is increased above 2 x ULN, total bilirubin should be differentiated into the direct and indirect reacting bilirubin. In any case, serum bilirubin should not exceed 1.6 mg/dL (27 μmol/L).
* History of renal trauma, glomerulonephritis, or patients with 1 kidney only, or a serum creatinine level exceeding 1.5 mg/dL (132.6 μmol/L).
* Screening total white blood cell (WBC) count < 3 000/μL, or platelets < 100 000/μL or neutrophils < 1 500/μL or hemoglobin < 8.5 g/dL (85 g/L).
* Active systemic infections during the last 2 weeks (exception: common cold) prior to registration.
* History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis according to local practice/guidelines) or a positive QuantiFERON TB-Gold test or TB-Spot Test (as indicated in Section 4.1 and Table 6-1). Patients with a positive test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active tuberculosis. If presence of latent tuberculosis is established then treatment according to local country guidelines must have been initiated.
* Known infection with human immunodeficiency virus, hepatitis B or hepatitis C at Screening or registration.
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 3 months, carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
* Use of Vitamin D containing supplements.
* Inability or unwillingness to undergo repeated venepuncture (e.g. because of poor tolerability or lack of access to veins).
* Patients who have received a live vaccine within 4 weeks prior to planned registration must be excluded.

Healthy Controls Inclusion Criteria:

* 10 healthy control blood samples.
* The healthy controls will be recruited from staff at the University of Liverpool or Aintree University hospitals and who are not taking nor have taken over the preceding 6 months, any immunosuppressive agent including systemic corticosteroids and whose health is otherwise good. There will be an equal balance of males to females. Matching to biologic or DMARD controls is not required. The healthy controls will provide one sample of blood for neutrophil studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in neutrophil apoptosis in PsA patients treated with Secukinumab at 12 months | 12 months
  Neutrophil apoptosis will be measured using flow-cytometry.
Change from baseline in neutrophil receptor expression in PsA patients treated with Secukinumab at 12 months | 12 months
  Neutrophil phenotype will be determine as percent of receptor expressing cells assessed by flow cytometry

SECONDARY OUTCOMES:
Change from baseline in neutrophil rate of phagocytosis in PsA patients treated with Secukinumab at 12 months | 12 months
  Neutrophil phagocytosis will be measured number of cells containing phagocytosis particles
Change from baseline in neutrophil chemotaxis in PsA patients treated with Secukinumab at 12 months | 12 months
  Neutrophil chemotaxis will be measured as the number of migrated neutrophil through cell inserts.
Change from baseline in Vitamin D receptor (VDR) expression in PsA patients treated with Secukinumab at 3 months | 3 months assessments from baseline
Change from baseline in Vitamin D receptor (VDR) expression in PsA patients treated with Secukinumab at 6 months | 6 months assessments from baseline
Change from baseline in Vitamin D receptor (VDR) expression in PsA patients treated with Secukinumab at 12 months | 12 months assessments from baseline
Change from baseline in quality of life in PsA patients treated with Secukinumab at 12 months using HAQ questionnaire | 12 months assessments from baseline
Change from baseline in quality of life in PsA patients treated with Secukinumab at 12 months using EQ5D questionnaire | 12 months assessments from baseline
Clinical response of psoriatic arthritis (ARC20) to treatment at 12 months | 12 months
Clinical response of psoriatic skin rash (PASI75) to treatment at 12 months | 12 months
Clinical response of of psoriatic Nail involvement (NAPSI) to treatment at 12 months | 12 months
Number of patients with treatment-related adverse events as assessed by MedDRA | 12 months
Number of patients with treatment-related serious adverse events as assessed by MedDRA | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Moots, MD PhD, Principal Investigator — University of Liverpool
Locations (1):
- Aintree University Hospitals NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
via publication
Supporting Information: CSR
Time Frame: Clinical trial results uploaded to EudraCT 12/03/2020